CLINICAL TRIAL: NCT03554109
Title: An Open-Label Randomized Phase 2 Trial Of The NANT NEOADJUVANT Triple-Negative Breast Cancer (TNBC) VACCINE VS Standard-Of-Care For The Neoadjuvant Treatment Of Subjects With TNBC
Brief Title: QUILT-3.057: NANT Neoadjuvant Triple- Negative Breast Cancer (TNBC) Vaccine
Acronym: TNBC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.057
Record Dates: First submitted 2018-05-25; First posted 2018-06-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2018-08

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Leucovorin; Fluorouracil; 130-nm albumin-bound paclitaxel; yeast-CEA vaccine; avelumab; ALT-803; Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Treatment will be administered in 2 phases, a neoadjuvant phase and a postoperative phase. For the experimental arm, subjects will receive treatment in the neoadjuvant phase for six 3-week cycles (ie, 18 weeks total). For the control arm, subjects will receive neoadjuvant treatment for a total of 16 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): NANT Neoadjuvant Triple Negative Breast Cancer Vaccine
  A combination of agents will be administered to subjects in this study:
  cyclophosphamide, 5-fluorouracil, leucovorin, nab-paclitaxel, avelumab, aldoxorubicin HCl, ALT-803, haNK, GI-4000, GI-6207, GI-6301, ETBX-011, ETBX-051 and ETBX-061
  Interventions: Drug: Leucovorin; Drug: 5-Fluorouracil; Drug: Aldoxorubicin HCl; Drug: nab-Paclitaxel; Biological: ETBX-011; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Drug: Avelumab; Biological: ALT-803; Biological: haNK; Drug: Cyclophosphamide
- Group B (Active Comparator): Standard treatment with a combination of doxorubicin, cyclophosphamide and paclitaxel.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin HCL; Drug: paclitaxel

INTERVENTIONS:
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  Arms: Group A
Drug: 5-Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Arms: Group A
Drug: Aldoxorubicin HCl — albumin-binding prodrug of doxorubicin HCl
  Arms: Group A
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
  Arms: Group A
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
  Arms: Group A
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
  Arms: Group A
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1[MUC1]
  Arms: Group A
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
  Arms: Group A
Biological: GI-6207 — CEA yeast vaccine
  Arms: Group A
Biological: GI-6301 — Brachyury yeast vaccine
  Arms: Group A
Drug: Avelumab — Avelumab
  Arms: Group A
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: Group A
Biological: haNK — NK-92 [CD16.158V, ER IL-2]
  Arms: Group A
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Doxorubicin HCL — Doxorubicin HCL
  Arms: Group B
Drug: paclitaxel — paclitaxel
  Arms: Group B

SUMMARY:
This is a randomized open-label phase 2 study to evaluate the efficacy and safety (as assessed by pCR) of the NANT Neoadjuvant TNBC Vaccine regimen (experimental arm) compared to the SoC dose-dense regimen of doxorubicin/cyclophosphamide followed by paclitaxel (control arm).

DETAILED DESCRIPTION:
Treatment will be administered in 2 phases, a neoadjuvant phase and a postoperative phase. The neoadjuvant phase will be 18 weeks for patients enrolled in the experimental arm and 16 weeks for those enrolled in the control arm.

Following the neoadjuvant phase, all subjects will undergo determination of their current response status and appropriate breast surgery and node dissection after which assessment for pCR will be conducted following completion of neoadjuvant systemic therapy. Pathologists interpreting surgical specimens for pCR assessment will be blinded to the treatment arm.

All subjects, regardless of whether or not they have achieved a pCR, will then enter the postoperative phase where they will receive adjuvant treatment. A small portion of the corresponding neoadjuvant therapy, either nab-paclitaxel or paclitaxel, will be administered as adjuvant treatment postoperatively. Adjuvant treatment will continue in the postoperative phase until the subject experiences unacceptable toxicity (not correctable with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically confirmed stage II or III TNBC. Subjects must be treatment naïve. TNBC is defined as breast cancer that lacks estrogen receptor (ER) and progesterone receptor (PgR) expression, and human epidermal growth factor receptor 2 (HER2) overexpression and/or amplification.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent FFPE tumor biopsy specimen and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator.
7. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
8. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, and autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease and ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) < 1,000 cells/mm^3.
   2. Platelet count < 75,000 cells/mm^3.
   3. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase (ALP) levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
7. Serious myocardial dysfunction defined by echocardiogram (ECHO) as absolute LVEF 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response Rate | 8 months
  Compare the efficacy of the NANT neoadjuvant TNBC Vaccine treatment vs standard-of-care (SoC) therapy as assessed by pathologic complete response (pCR) rate in the breast and axilla.

SECONDARY OUTCOMES:
Evaluation of safety as determined by incidence or treatment-emergent adverse events | 36 months
  Incidence of treatment -emergent adverse events
Evaluate additional measures of efficacy by event-free survival | 36 months
  Time from randomization to first occurrence of advancement of disease
Overall survival | 36 months
  Time from date of first treatment to death from any cause
Locoregional relapse | 36 months
  Presence of any disease recurrence, including location
Distant metastatic rates at 1 year | 36 months
  Number of patients with a metastatic lesion

OTHER OUTCOMES:
Quality of life by patient-reported outcomes | 36 months
  Score on FACT-B QoL Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No